CLINICAL TRIAL: NCT06070064
Title: Effects of Trap and Reggaeton Music on Movement Velocity, Power and Muscular Endurance in the Lower Limbs of Physically Active Women
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Seville (Other)
Responsible Party: Principal Investigator, Jimenez-Roldan Manuel Jesus, Principal Investigator, University of Seville
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Other
Other Study IDs: Trap_Strength_women
Record Dates: First submitted 2023-09-05; First posted 2023-10-06 (Actual); Last update posted 2023-10-06 (Actual); Status verified 2023-09

CONDITIONS: Female; Sports; Muscle; Exercise
MeSH Terms: conditions — Motor Activity

STUDY DESIGN:
Intervention Model Description: The investigators intend to conduct an experimental trial with a randomised crossover design in 12 participants physically active young women adults with strength training experience aged 18-30 years.
  The study will be conducted in the laboratory of Physical Activity and Sport Sciences of the University School of Osuna.
  In this way, at the end of the study will have contrasted scientific information on the effects of music on the following variables of speed of execution in the back squat exercise.
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: Participants will complete two additional randomised, counterbalanced visits, each with a different condition: (a) Music (b) Non-Music.
  To ensure participants are blinded, they will be given detailed instructions on the Study Information Sheet, indicating that they will come to the laboratory to perform the assessment tests in different environmental conditions that will not impact on their health status.
  which will not affect their health status. Experimental measurements will be taken in the morning, at the same time of day (±0.5 h) for each individual, to standardise the influence of circadian rhythm, at a temperature of 23°C (±1°C).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Music (Experimental): The "music" group will carry out an initial familiarisation session of the main study variables. Subsequently, through an incremental test, MR will be evaluated through the control of execution speed.
  The heaviest load at which each participant could correctly lift with full knee extension shall be considered as their 1RM.
  For lighter loads (average speed> 1.0 m-s-1), there will be 3 attempts per load.There shall be two attempts with medium loads(0.50 m-s-1 ≥ average speed ≤ 1.0 m-s-1); and only one for close to maximum loads (average speed < 0.50 m-s-1).
  After the first 1RM visit described above, participants will complete two additional random counterbalanced visits, each with a different condition.
  The music group started the whole evaluation process with the music conditioning factor present. After completion of the measurements and the necessary rest time, the measurement was repeated in the non-music condition.
  Interventions: Other: Effect of music on the manifestation of strength
- Non-music (Experimental): The "non-music" group developed the same protocol but started the measurements without the presence of music.
  Interventions: Other: Effect of music on the manifestation of strength

INTERVENTIONS:
Other: Effect of music on the manifestation of strength — After the first 1RM visit, described above, each participant will complete 2 additional randomised, counterbalanced visits, each with one condition: Music (MUS) and No Music (No-MUS). The participants will be instructed to attend the laboratory to perform the screening test in different environmental conditions that do not impact on their health status.
  During the MUS session, participants will perform a back squat test and a CJM test while listening to music. The chosen songs will be at least 120 beats per minute (BPM) 15. The tempo of the music for each of the tracks will be calculated using bpm software (Tangerine!v.1.4). The music will be played using an iPhone X (Apple Inc., Cupertino, CA, USA) connected to a portable speaker (Sony MHC-V02, Sony Co., Tokyo, Japan). The sound intensity will be adjusted and standardised for all participants to 75 dB (at ear level) using the Decibel X-dBA sound level meter. Trap and reggaeton music will be played before, during and after the test.

SUMMARY:
The influence of music on movement velocity and power during strength training have been poorly investigated, and specifically in women there is no evidence of an increase in strength performance due to the influence of music.

Hypothesis: Listening to trap or reggaeton music will improve jumping ability, as well as movement velocity and power, muscular endurance, motivation and perception of effort in trained women during the performance of back-squats.

DETAILED DESCRIPTION:
The investigators pretend to conduct an experimental trial with a randomised crossover design in 28 participants physically active young adults with strength training experience aged 18-30 years. The study will be conducted in the laboratory of Physical Activity and Sport Sciences of the University School of Osuna.

In this way, at the end of the study the investigatos will have contrasted scientific information on the effects of music on the following variables of speed of execution in the back squat exercise.

back.

ELIGIBILITY:
Inclusion Criteria:

* more than 6 months performing strength training programmes
* familiarity with back squat exercises
* no consumption of any type of nutritional supplement or anabolic substances in the three months prior to or during the same study period; v) absence of musculoskeletal injuries that may interfere with the exercise protocol during the investigation
* absence of musculoskeletal injuries that may interfere with the exercise protocol during the investigation
* normal hearing ability

Exclusion Criteria:

* in addition to the above inclusion criteria, the following shall be excluded from the study participants who do not sign the informed consent form.

Ages: 18 Years to 30 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes
Enrollment: 14 (Actual)
Dates: Start 2023-06-01 (Actual); Primary Completion 2023-06-15 (Actual); Study Completion 2023-06-30 (Actual)

PRIMARY OUTCOMES:
Jumping Ability (CMJ Test) | up to 4 weeks
  Day 1 (First situation: Music or non-music) Before assessing the participants, a warm-up with familiarisation with the CMJ will be performed. This will be followed by a short specific warm-up of 5 jumps.
  After a couple of minutes of rest, the test will be performed with 3 CMJs. The jumping technique consists of a flexion-extension of hips and knees at the highest possible speed to jump as high as possible; the knee angle at maximum flexion should be close to 90° and then return to the starting position. Participants will be encouraged to perform the maximum jump height in the concentric phase of each repetition to ensure maximum muscular strength.
  So, this test shall be performed at baseline and after maximal effort.
  Day 2: Second situation: The same protocol but in the other situación allocated.
Movement Velocity and Power in Back-Squat at 50% and 75% 1RM (Mean and Peak Measurements) | Up to 4 weeks
  Day 1 (First situation: Music or non-music)
  Each participant will be given the same warm-up protocol as for assessing 1RM.
  After 3 min rest: Two back squats will be performed using a Smith machine while movement speed and power will be measured.
  The first test will consist of 2 repetitions at 50% of 1RM.
  After 3 minutes rest: The second test will be performed. It will consist of 2 repetitions at 75% of 1RM.
  Both tests shall be performed at maximum speed. Participants shall be encouraged to perform the best possible effort in the concentric phase of each repetition to ensure maximum muscular strength. The average speed in m/s will be recorded for both repetitions, as well as the maximum speed of both squats (at 50% and 75% of 1RM). The velocity of movement will be monitored by the researchers using a validated linear position transducer.
  Day 2: Second situation: The same protocol but in the other situación allocated.
Muscular Endurance | Up to 4 weeks
  Day 1 (First situation: Music or non-music)
  After 3 minutes rest, a test shall be performed to calculate the maximum number or repetitions to concentric failure at 75% of 1RM.
  Day 2: Second situation: The same protocol but in the other situación allocated.
Participants motivation through an Analogic Visual Scale (AVS) | Up to 4 weeks
  Day 1 (First situation: Music or non-music)
  The AVS will consist of a 100 mm straight line where 0 mm indicates "no motivation", while 100 mm indicates "extremely motivated". Participants will mark on the line how motivated they feel during the exercise. Researchers will then record the distance between 0 mm and the mark participants place on the line.
  Day 2: Second situation: the same protocol but in the other situación allocated.
Participants Perceived Effort | Up to 4 weeks
  Day 1 (First situation: Music or non-music)
  As soon as participants complete the muscular endurance test, perceived exertion will be assessed on a scale of 0 (minimun) to 10 (maximum). The answers given will be recorded by the researchers.
  Day 2: Second situation: the same protocol but in the other situación allocated.

CONTACTS AND LOCATIONS:
Locations (1):
- Education Faculty, Seville, Spain

IPD SHARING:
Plan to Share IPD: No